CLINICAL TRIAL: NCT00937157
Title: Comparison of Standard 1.5 Versus 3T Optimized Protocols in Patients Treated With Glatiramer Acetate. A Conventional and Non-conventional MRI Study
Brief Title: Comparison of 1.5T vs. 3T Protocols After Treatment With Glatiramer Acetate (GA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Teva Neuroscience, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Professor of Neurology, University at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BNAC/GA/01
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Results first posted 2014-12-09 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
Keywords: Inflammation; Multiple Sclerosis; Glatiramer Acetate; Gd enhancing lesions; 1.5T protocol; 3T protocol; Magnetization transfer imaging (MTI); Lesion activity analysis; Copaxone
MeSH Terms: conditions — Multiple Sclerosis; Inflammation | interventions — Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Patients diagnosed with multiple sclerosis who have the presence of at least 1 or more Gd enhancing lesions and/or acute relapse.
  Interventions: Drug: Copaxone

INTERVENTIONS:
Drug: Copaxone — 12 MS patients will be enrolled on GA (Copaxone®) monotherapy (20mg/day sc). Initial intravenous steroid treatment will be given on day 0. 1.5T and 3T scans will be obtained and according to the following schedule: 1 gm Solumedrol i.v. daily for three days. Intravenous steroids will be also allowed for treatment of MS attacks according to the following schedule: 1 gm Solumedrol i.v. daily for three days.
  Other Names: Glatiramer acetate

SUMMARY:
This study will:

* Explore whether GA decreases inflammation more on the 3T optimized protocol when compared to the 1.5T standard protocol.

  * Compare whether the decrease in the cumulative number of Gd-enhancing lesions significantly differs between pre-treatment (day 0) and post-treatment (12 months) using 1.5T standard and 3T optimized protocols.
* Investigate the correlation between MTR and the cumulative number and volume of Gd enhancing lesions on 1.5T standard and 3T optimized protocols in patients treated with GA.

This study suggests that GA may favorably affect early events in lesion formation, in addition to exerting more transient beneficial effects on established areas of inflammation and demyelination, and that this effect may be observed only with the 3T optimized protocol.

DETAILED DESCRIPTION:
Interferon-β (IFN- β) and glatiramer acetate (GA) are the two main groups of drugs used in the treatment of multiple sclerosis (MS). Notably, while both ultimately decrease central nervous system (CNS) inflammation, they do so by very different mechanisms. Therefore, use of 1.5T MRI, triple dose of Gd, delay of scanning time for 20-30 min after Gd injection, and application of off-resonance saturated MT pulse may increase the ability to detect Gd lesions by approximately 120% when compared to 1.5T single dose MRI protocol. The 3T standard protocol may increase the ability to detect Gd enhancing lesions by 40-50% when compared to the 1.5T standard protocol. This may indicate that the 3T optimized protocol may increase the ability for Gd lesion detection by approximately 150-180%, when compared to the 1.5T standard protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with clinically definite MS according to the McDonald criteria
* Have a Gd enhancing lesion using 1.5T standard protocol and/or an acute relapse
* Age 18-65
* Have a relapsing-remitting (RR) disease course or clinically isolated syndrome (CIS) with high risk of conversion to clinically definite (CD) MS (presence of >9 T2 lesions in addition to 1 Gd lesion)
* Have EDSS scores less than or equal to 5.5
* Have disease duration of 3 months to 30 years
* None of the exclusion criteria

Exclusion Criteria:

* Previous immunomodulatory or immunosuppressant treatment during the 30 days prior to day 0 of the study with the following agents (e.g., IFN-β, GA, mitoxantrone, cyclophosphamide, cladribine, fludarabine, cyclosporine, total body, azathioprine, methotrexate, IVIG, cellcept, natalizumab, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, MD, PhD, Principal Investigator — University at Buffalo
Locations (1):
- Jacobs Neurological Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from the pool of relapsing-remitting multiple sclerosis patients (RRMS) at the Jacob's Neurological Institute (JNI) was open for approximately one year.
Pre-assignment Details: All enrolled patients had to meet all inclusion criteria and no exclusion criteria. Patients were to be 18-65 years of age, have a disease duration of 3months to 20 years, be diagnosed with RRMS according to McDonald criteria, one enhancing lesion 30 days prior to screening and an EDSS score equal to or below 5.5.
Groups:
- RRMS Patients With >=1 GdE Lesion or Acute Relapse: Patients diagnosed with multiple sclerosis who have the presence of at least 1 or more Gd enhancing lesions and/or acute relapse.
  Copaxone: 12 MS patients were enrolled on GA (Copaxone®) monotherapy (20mg/day sc). Initial intravenous steroid treatment was given on day 0. 1.5T and 3T scans were obtained according to the following schedule: 1 gm Solumedrol i.v. daily for three days. Intravenous steroids were also allowed for treatment of MS attacks according to the following schedule: 1 gm Solumedrol i.v. daily for three days.
Period: Overall Study
Arm/Group | RRMS Patients With >=1 GdE Lesion or Acute Relapse
Started | 12
Completed | 8
Not Completed | 4
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Groups:
- Patients Diagnosed With Multiple Sclerosis Who Have the Presen: Copaxone: 12 MS patients will be enrolled on GA (Copaxone®) monotherapy (20mg/day sc). Initial intravenous steroid treatment will be given on day 0. 1.5T and 3T scans will be obtained and according to the following schedule: 1 gm Solumedrol i.v. daily for three days. Intravenous steroids will be also allowed for treatment of MS attacks according to the following schedule: 1 gm Solumedrol i.v. daily for three days.
Arm/Group | Patients Diagnosed With Multiple Sclerosis Who Have the Presen
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (7.823)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: A Change in the Cumulative Number of Gd Enhancing Lesions Using a 3T Protocol.
Time Frame: Change from baseline at 180 days and change from baseline at 360 days
Population: Of the 12 RRMS patients enrolled, only the 8 who completed days 180 and 360 were analyzed. There was no imputation used.
Measure: Mean (Standard Deviation); unit: GAD lesions (number of)
Units Other Than Participants: GAD lesions
Arm/Group | Patients Diagnosed With Multiple Sclerosis Who Have the Presen
Number analyzed (Participants) | 8
Number analyzed (GAD lesions) | 16
GAD lesions (number of)
  GAD lesions from 0-180 | -3.7 (5.8)
  GAD lesion from 0-360 | -3.6 (4.2)

ADVERSE EVENTS:
Arm/Group | RRMS Patients With >=1 GdE Lesion or Acute Relapse
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No